CLINICAL TRIAL: NCT00575627
Title: Treatment of Chronic Hepatitis C Patients With Persistently Normal Alanine Aminotransferase Levels With Peginterferon α-2a (40 kDa) Plus Ribavirin
Brief Title: Pegylated-Interferon and Ribavirin in Hepatitis C Patients With Persistently Normal Alanine Aminotransferase Levels
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Prof Mario Rizzetto - Dipartimento di GastroEpatologia - Università degli Studi di Torino, Università degli Studi di Torino
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: pNNALTHCV; NNALT
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis C; persistently normal ALT; pNNALT; Theraphy for Hepatitis C; Pegylated Interferon; Combined therapy
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (No Intervention)
- 1 (Experimental): Drug: peginterferon α-2a (40 kDa) plus ribavirin for 24-48 weeks
  Interventions: Drug: Peg-Interferon alpha2a plus Ribavirin

INTERVENTIONS:
Drug: Peg-Interferon alpha2a plus Ribavirin — Peg-Interferon alpha2a: 180 micrograms per week Ribavirin:100-1200 mg/daily
  Arms: 1

SUMMARY:
Patients with chronic hepatitis C with persistently normal alanine aminotransferase (ALT) levels have been generally excluded from treatment, because the strong conviction that normal ALT would be synonymous of absence of liver damage. However, recent studies have demonstrated marked liver fibrosis, including cirrhosis, in patients with HCV and persistently normal ALT levels. Up to now, just a sigle randomized, controlled, multicenter study was lead to evaluate the efficacy and safety of combined therapy in patients with chronic hepatitis C and persistently normal serum ALT levels. Aim of our study is evaluate the efficacy of treatment and the outcome of treated patients compared with a control group of untreated patients.

ELIGIBILITY:
Inclusion Criteria:

* Serologic evidence of chronic hepatitis C infection (repeatedly HCV-RNA positive) with persistent normal ALT levels documented on at least 3 occasions, in the last 18 months before screening.
* Fibroscan performed in the last 3 months
* Compensated liver disease, Child Pugh score <7
* Serum HCV-RNA >615 IU/mL
* Patients who are naïve to any hepatitis C therapy (i.e. have not been previously treated with an interferon or with IFN plus ribavirin)
* No clinical or radiological evidence of hepatocellular carcinoma and a serum AFP <100 ng/mL within 2 months of randomisation
* Negative urine or blood pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of study drug
* All fertile males and females receiving ribavirin must be using two forms of effective contraception during treatment and during the 6 months after treatment end

Exclusion Criteria:

* Women with ongoing pregnancy or breast feeding
* History or other evidence of bleeding from oesophageal varices or other conditions consistent with decompensated liver disease (Child Pugh B or C)
* Therapy with any systemic anti-viral, anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) £6 months prior to the first dose of study drug
* History or other evidence of a medical condition associated with chronic liver disease other than HCV (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures)
* Neutrophil count <1500 cells/mm3 or platelet count <90,000 cells/mm3 at screening
* Serum creatinine level >1.5 times the upper limit of normal at screening
* Evidence of current severe psychiatric disease, especially depression within one year of study entry. Severe psychiatric disease is defined as treatment with an antidepressant medication or a major tranquilizer at therapeutic doses for major depression or psychosis, respectively, within 12 months prior to study entry. Patients with a previous history of the following: a suicidal attempt, hospitalization for psychiatric disease, or a period of disability due to a psychiatric disease should be evaluated by a qualified Psychiatrist for study suitability prior to enrolment.
* History of a severe seizure disorder or current anticonvulsant use History of immunologically mediated disease, chronic pulmonary disease associated with functional limitation, severe cardiac disease, major organ transplantation or other evidence of severe illness, malignancy, or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study
* History of thyroid disease poorly controlled on prescribed medications, elevated thyroid stimulating hormone (TSH) concentrations with elevation of antibodies to thyroid peroxidase and any clinical manifestations of thyroid disease
* Evidence of severe retinopathy (e.g. CMV retinitis, macula degeneration)
* Evidence of drug abuse (including excessive alcohol consumption) within 6 months of study entry
* Inability or unwillingness to provide informed consent or abide by the requirements of the study
* Male partners of women who are pregnant
* Hgb <12 g/dL in women or <13 g/dL in men at screening
* Any patient with an increased baseline risk for anemia (e.g. thalassemia, spherocytosis, history of GI bleeding, etc) or for whom anemia would be medically problematic
* Patients with documented or presumed coronary artery disease or cerebrovascular disease should not be enrolled if, in the judgment of the investigator, an acute decrease in hemoglobin by up to 4 g/dL (as may be seen with ribavirin therapy) would not be well-tolerated

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-09 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of treatment and the outcome of treated patients compared with a control group of untreated patients. | 48-72 weeks

SECONDARY OUTCOMES:
evaluation of liver fibrosis by Fibroscan after 48-72 weeks of inclusion | 48-72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rizzetto Mario, Principal Investigator — Università degli Studi di Torino - Azienda Ospedaliera San Giovanni Battista di Torino, Molinette,
Locations (1):
- Università degli Studi di Torino - Azienda Ospedaliera San Giovanni Battista di Torino, Molinette,, Torino, Italy